CLINICAL TRIAL: NCT06889805
Title: Universal Screening for Hepatitis Delta Virus (HDV) in Individuals Living with HIV/HBV Coinfection and HBV-related HCC
Brief Title: HDV Screening Study
Status: Recruiting | Type: Observational
Sponsor: Grace Lai Hung Wong (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Grace Lai Hung Wong, Professor, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Other Study IDs: SPEARHEAD 2024
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis D Virus Infection
Keywords: HDV
MeSH Terms: conditions — Hepatitis D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a territory-wide cross-sectional study of all individuals living with HIV/HBV coinfection and HBV-related HCC.

DETAILED DESCRIPTION:
Chronic hepatitis B virus (HBV) infection remains endemic in Hong Kong with an estimated prevalence of 6.2% in the recent Population Health Survey 2020-2022.1 The estimated prevalence of chronic HBV infection among individuals living with HIV is 8%.2 Yet, no data are available concerning the disease burden of hepatitis delta virus (HDV) among individuals living with HIV/HBV coinfection.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with HIV infection, i.e. anti-HIV or HIV RNA positive; AND
2. Individuals with chronic hepatitis B, i.e. hepatitis B surface antigen (HBsAg) or HBV DNA positive for two times at least 6 months apart; AND
3. Aged 18 years old or above.
4. Written or verbal consent obtained

Exclusion Criteria:

1. Refusal to consent
2. Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals living with HIV/HBV coinfection and HBV-related HCC
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2028-08-17 (Estimated); Study Completion 2029-02-17 (Estimated)

PRIMARY OUTCOMES:
Rate of positive anti-HDV | at screening
  Primary endpoint is seroprevalence rate of positive anti-HDV

SECONDARY OUTCOMES:
Prevalence rate of detectable HDV RNA | at screening
  Prevalence rate of detectable HDV RNA
Prevalence rate of compensated advanced chronic liver disease | at screening
  Prevalence rate of compensated advanced chronic liver disease (cACLD) defined as a liver stiffness measurement above 10.0 kPa

CONTACTS AND LOCATIONS:
Overall Officials: Lai Hung Grace Wong, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lai JC, Wong GL, Wong VW, Yip TC. Unmet need in screening for hepatitis D virus: Time to take action. J Hepatol. 2024 Jun;80(6):e277-e278. doi: 10.1016/j.jhep.2023.12.006. Epub 2023 Dec 16. No abstract available. PMID 38110005
- [Background] Lui GC, Wong GL, Yang HC, Sheng WH, Lee SH. Current practice and recommendations for management of hepatitis B virus in people living with HIV in Asia. HIV Med. 2023 Oct;24(10):1035-1044. doi: 10.1111/hiv.13545. Epub 2023 Sep 21. PMID 37735948